CLINICAL TRIAL: NCT04744389
Title: Optimization of an Evidence-based Organizational Model of Liver and Pancreas Transplant Using Cardiac Death Donors: a Pilot, Prospective, Randomized, Multicenter Study for the Comparison of Hypothermic Versus Normothermic Ex-vivo Preservation.
Brief Title: Comparison of Hypothermic Versus Normothermic Ex-vivo Preservation.
Acronym: DCDNet
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Collaborators: Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy (Other Government); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Davide Ghinolfi, Principal Investigator, Azienda Ospedaliero, Universitaria Pisana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D52F20000740002
Record Dates: First submitted 2021-01-18; First posted 2021-02-09 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: End Stage Liver DIsease
Keywords: ex-situ perfusion; organ preservation; normothermic perfusion; hypothermic perfusion
MeSH Terms: conditions — End Stage Liver Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypothermic Machine Perfusion (Experimental): uDCD and cDCD after Normothermic Regional Perfusion matching the inclusion criteria, ECD matching the inclusion criteria, uDCD and cDCD exceeding the inclusion criteria.
  Interventions: Device: Hypothermic Machine Perfusion
- Normothermic Machine Perfusion (Experimental): uDCD and cDCD after Normothermic Regional Perfusion matching the inclusion criteria, ECD matching the inclusion criteria, uDCD and cDCD exceeding the inclusion criteria.
  Interventions: Device: Normothermic Machine Perfusion

INTERVENTIONS:
Device: Hypothermic Machine Perfusion — The perfusion system was primed with 4 L of Belzer machine perfusion solution University of Wisconsin Machine Perfusion Solution (Bridge for Life, Ltd., Columbia, SC). The arterial and portal pressures were set at 25 mm Hg with a flow and at 3-4 mm Hg with a continuous flow, respectively. The oxygen flow was set at 0.25 L/minute. The target liver temperature was between 4°C and 10°C.
  Other Names: Hypothermic machine perfusion (HMP)
  Arms: Hypothermic Machine Perfusion
Device: Normothermic Machine Perfusion — Grafts were perfused at 37°C in an OR next to the transplant OR and under medical supervision using a blood-based perfusate. Initial perfusate temperature was set at 20°C and raised by 1°C every 2 minutes. Oxygenation was provided by an anesthesia ventilator initially set at 4 L/minute with 30% fraction of inspired oxygen, and later adjusted based on perfusate pH, partial pressure of oxygen, and partial pressure of carbon dioxide. Blood gas analyses were drawn every 20 minutes during the first hour and every 30 minutes thereafter with the aim to maintain a physiological pH and ionogram result, and a partial pressure of oxygen between 200 and 250 mm Hg. Perfusate glucose, transaminases, and lactate were measured during NMP as were bile production and quality (pH, sodium, glycemia, lactate, and HCO3)
  Other Names: Normothermic machine perfusion (NMP)
  Arms: Normothermic Machine Perfusion

SUMMARY:
Study groups:

The study is a multicenter (Pisa and Milan), prospective, randomized study comparing D-HOPE (HMP) vs NMP in DCD and ECD-DBD (extended criteria brain-dead donors). Once a DCD or a DBD with extended criteria (ECD-DBD) meets the inclusion criteria, they are randomized as follow:

1. 20 liver grafts from DCD after normothermic regional perfusion (NRP) matching the inclusion criteria are randomized 1:1 to hypothermic machine perfusion (HMP) vs normothermic machine perfusion (NMP) and then transplanted.
2. 40 liver grafts from ECD-DBD matching the inclusion criteria are randomized 1:1 to hypothermic machine perfusion (HMP) vs normothermic machine perfusion (NMP) and then transplanted

DETAILED DESCRIPTION:
The persistent mismatch between patients waiting for a liver transplant (LT) and grafts availability promoted the use of donation after circulatory death (DCD). Italian law requires 20 minutes of continous flatline electrocardiogram to declared individual's circulatory death and such a long period of warm ischemia time forced the development of protocols using abdominal normothermic regional perfusion (NRP) followed by ex-vivo graft reperfusion by means of machine perfusion technology (MP) for its potential to minimize ischemia/reperfusion damage and promote organ repair and reconditioning prior to transplantation. An extensive evaluation of all DCD donors might increase donation rate by 30%, but, while kidney transplant from DCD donors is well implemented, no definitive data exist on the optimal use of NRP and MP in liver and pancreas transplantation and an organizational model is far to be implemented. Moreover, a randomized trial comparing hypothermic vs normothermic ex-vivo perfusion has never been performed. The proposed project will perform a pilot, open, randomized, prospective trials to evaluate the sequential use of NRP followed by ex-vivo MP (hypothermic (HMP) vs normothermic (NMP)) by measuring several indicators of organ damage and recovery with the target to set up the optimal organizational model for DCD donation:

1. Twenty LT from DCD donors after NRP (considered transplantable for the acceptance criteria in use) will be randomized 1:1 to ex-vivo HMP or NMP (multicenter study together with the center in Milan)
2. 40 liver grafts from ECD-DBD matching the inclusion criteria are randomized 1:1 to hypothermic machine perfusion (HMP) vs normothermic machine perfusion (NMP) and then transplanted To assess organ damage and repair capacity, the following investigations will be performed: -biomarkers of apoptosis, necrosis, innate-mediated inflammation and its resolution, angiogenesis and thrombosis during NRP -circulating biomarkers indicating damage, proliferation, angiogenetic and tissue remodelling factors; a targeted-metabolomic and lipidomic profiling during ex-vivo HMP or NMP in the perfusate and on blood samples in the peri and post-operative period; bile composition on graft subjected to NMP. Evaluation of necrosis, apoptosis and proliferation, immunohistochemical analysis, a targeted-metabolomic and lipidomic profiling, ATP measurement, and electronic microscopy investigations will be performed on liver tissue and bile duct biopsies after NRP, before and after ex-vivo reperfusion, and immediately after reperfusion in the recipient (only for transplantable grafts) Based on the collected data a new algorithm of organ evaluation, procurement, preservation and reconditioning will be formulated and disseminated.

ELIGIBILITY:
GRAFT:

Inclusion criteria:

DCD:

* no absolute contraindications as per Italian National Transplant center (CNT)
* donor age ≤70 years
* witnessed and documented cardiac arrest
* macro-vescicular steatosis <30% at liver biopsy
* necrosis <5% at liver biopsy
* fibrosis <2 as per Ishak's score at liver biopsy
* arteriolar thickening <60% at liver biopsy
* WIT ≤160 minutes
* ALT <1000 UI/L during NRP
* downward trend lactate during NRP

DBD:

* no absolute contraindications as per Italian National Transplant center (CNT)
* donor age > 70 years
* macro-steatosis between 30 and 50% at liver biopsy

Exclusion criteria:

DCD:

* absolute contraindications as per Italian National Transplant center (CNT)
* donor age >70 years
* macro-vescicular steatosis >30% at liver biopsy
* necrosis >5% at liver biopsy
* fibrosis >2 as per Ishak's score at liver biopsy
* severe macroangiopathy (arteriolar thickening >60% at liver biopsy)
* WIT >160 minutes
* ALT >1000 UI/L during NRP
* uptrend lactate during NRP

DBD:

* absolute contraindications as per Italian National Transplant center (CNT)
* donor age < 70 years
* macro-steatosis between > 50% at liver biopsy

RECIPIENTS

Inclusion criteria:

* Subject must be greater than or equal to 18 years of age.
* Subject with end-stage liver disease who is actively listed for primary liver transplantation
* Subject, or a legally authorized representative, has given informed consent to participate in the study

Exclusion criteria:

* Subject is currently listed as a UNOS status 1A.
* Subject is requiring oxygen therapy via ventilator/respiratory support.
* Subject is planned to undergo simultaneous solid organ transplant.
* Subject is pregnant at the time of transplant.
* Subject MELD score 25 or higher
* Subject receives re-transplantation of liver.
* Any medical conditions contro-indicating the use of DCD grafts at transplant surgeon/hepatologist evaluation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Rate of graft loss | at 6 months postoperatively
  Death of patient, relisting or Retransplantation. Composite Outcome
Rate of Ischemic Type Biliary Lesions (ITBL) | at 6 months postoperatively
  ITBL as assessed by MRI / MRCP. Composite Outcome

SECONDARY OUTCOMES:
1-year graft survival | 1-year postoperatively
1-year patients survival | 1-year postoperatively
level of BCL-2/BAX at the liver histology | after 2 hours of perfusion
  BCL-2/BAX is members of the Bcl-2 family of regulator proteins that regulate cell death and correlates with graft loss
level of Soluble Keratin 18 in the perfusate | after 2 hours of perfusion
  Soluble Keratin 18 is a marker of necrosis and apoptosis and correlates with graft loss
level of HMGB1in the perfusate | after 2 hours of perfusion
  HMGB1 Acts as danger associated molecular pattern (DAMP) molecule that amplifies immune responses during tissue injury and correlates with graft loss

CONTACTS AND LOCATIONS:
Locations (1):
- UO Chirurgia Epatica e del Trapianto di Fegato, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ghinolfi D, Rreka E, De Tata V, Franzini M, Pezzati D, Fierabracci V, Masini M, Cacciatoinsilla A, Bindi ML, Marselli L, Mazzotti V, Morganti R, Marchetti P, Biancofiore G, Campani D, Paolicchi A, De Simone P. Pilot, Open, Randomized, Prospective Trial for Normothermic Machine Perfusion Evaluation in Liver Transplantation From Older Donors. Liver Transpl. 2019 Mar;25(3):436-449. doi: 10.1002/lt.25362. PMID 30362649
- [Background] Ghinolfi D, Dondossola D, Rreka E, Lonati C, Pezzati D, Cacciatoinsilla A, Kersik A, Lazzeri C, Zanella A, Peris A, Maggioni M, Biancofiore G, Reggiani P, Morganti R, De Simone P, Rossi G. Sequential Use of Normothermic Regional and Ex Situ Machine Perfusion in Donation After Circulatory Death Liver Transplant. Liver Transpl. 2021 Feb;27(3):385-402. doi: 10.1002/lt.25899. Epub 2020 Nov 8. PMID 32949117
- [Derived] Lazzeri C, Ghinolfi D, Santini LE, Procissi APO, Cultrera D, Peris A. Improved Utilization Rate in Solid Organ Donors >/=80 Years: The 7-Year Tuscany Experience. Clin Transplant. 2025 Apr;39(4):e70142. doi: 10.1111/ctr.70142. PMID 40145941
- [Derived] Tingle SJ, Thompson ER, Figueiredo RS, Moir JA, Goodfellow M, Talbot D, Wilson CH. Normothermic and hypothermic machine perfusion preservation versus static cold storage for deceased donor kidney transplantation. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD011671. doi: 10.1002/14651858.CD011671.pub3. PMID 38979743